CLINICAL TRIAL: NCT04282304
Title: Randomised Trial of Comprehensive, Intensive, On-site Behavioural Lifestyle Intervention Versus Usual Care During the Preoperative Preparation for Bariatric Surgery
Brief Title: Randomised Trial of Intensive Behavioral Lifestyle Intervention Versus Usual Preparation for Bariatric Surgery
Acronym: PICO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Premature termination due to lack of inclusion. Behavioral preparation is perceived as too restrictive by patients. Furthermore, the Covid and post-covid period has drastically restricted the possibilities of support for behavioral preparation.
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-006
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Morbid Obesity
Keywords: Behavioral intervention; Severe obesity; Weight loss; Bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Other): The patients in this arm will have usual care during preoperative period, bariatric surgery and follow-up.
  Interventions: Behavioral: Preoperative usual care
- UGECAM (Experimental): During the preoperative period, the patients in this arm will have usual care and a 4 weeks intensive, comprehensive behavioral lifestyle intervention. They will then have usual bariatric surgery and follow-up.
  Interventions: Behavioral: Preoperative intensive behavioral lifestyle intervention

INTERVENTIONS:
Behavioral: Preoperative usual care — Usual care during the preoperative preparation for bariatric surgery consists of:
  * Endocrinologist work-up and follow-up, with at least 2 consultations;
  * Dietary advice, provided during the endocrine consultation or dietician consultation
  * Psychological counselling with the patient's usual psychiatrist (at least 2 consultations
  * Physical activity and nutrition are encouraged, but entrusted to the patient's freedom of choice. Weight loss, or at least, weight stabilization, is recommended before the surgery, without initiating a specific behavioural procedure.
  Arms: Usual Care
Behavioral: Preoperative intensive behavioral lifestyle intervention — The intensive behavioral lifestyle intervention program takes place over 4 weeks of 5 days. It includes:
  * Rehabilitation to physical exercise every morning
  * Therapeutic cooking sessions; during these sessions, the patients prepare the day's meals under the supervision of a nutritionist
  * Psychological counselling
  * One swimming session per week
  * One relaxation session
  * Regular physical activity (aerobics, work-up)
  * Individual entertainment with the physiotherapist physician and discussion groups
  * Weight, BMI and waist circumference control at the end of each week.
  Arms: UGECAM

SUMMARY:
Prospective randomized clinical trial aiming to compare a comprehensive, intensive behavioral lifestyle intervention and usual care during the preoperative preparation to bariatric surgery, with primary outcome on excess weight loss and secondary outcomes on patient's physical status, quality of life, comorbidity and technical difficulty of the surgery.

DETAILED DESCRIPTION:
Obesity is a complex, multifactorial pathology that has major public health importance. Lifestyle modification is the cornerstone of all obesity treatments, including surgery. Throughout the non-surgical treatment options, high-intensity, on-site comprehensive lifestyle intervention has demonstrated the best efficacy in obtaining weight loss, but with a risk of progressive weight regain, after 6 months (1). In obese adults, bariatric surgery produces greater weight loss and weight loss maintenance than the conventional medical treatment and lifestyle intervention (1).

There is no consensus on whether combining these two approaches (i.e. high-intensity, on-site comprehensive lifestyle intervention and bariatric surgery) results in enhanced weight loss or more sustainable outcomes. The present randomized trial aims to answer this question.

Patients preparing for bariatric surgery will be randomized between two groups. The first group will receive the usual care as recommended by the French Health Authority ("Haute Autorité de santé"), including 6 months of endocrine and nutritional follow-up and educational intervention. The second group will receive a high-intensity, 4 weeks on-site comprehensive lifestyle intervention, including prescription of a moderately reduced-calorie diet, a program of increased physical activity, and behavioral management. The patients from both groups will then be operated on and followed for at least 2 years. Complete work-up, including clinical examination, comorbidity assessment, MRI of the liver, thigh and abdominal fat, 6 minutes' walk test, quality of life questionnaires will be performed at the begging of the follow-up, after the preparation (usual care or intensive) and 2 years after surgery. Clinical and biological assessment will be performed regularly after surgery, and technical details from the bariatric interventions will be analyzed in order to assess the eventual facilitation of the gestures in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a BMI (Body Mass Index) of 40 or BMI of 35 with associated comorbidity and who desires obesity surgery
* Patient agreeing to participate in the study, including the 2 years follow-up
* Patient accepting the constraints of the study related to the group to which he/she will be assigned as a result of randomization (availability to his work, his family, etc.)
* Patient able to receive and to understand the study information and to give written informed consent
* Patient affiliated with the French social security system

Exclusion Criteria:

* Patient with a BMI of more than 60
* Patient with contraindication to laparoscopic obesity surgery
* Patient already operated on for obesity
* Patient with a history of major abdominal surgery
* Patient with contraindications to MRI:

  * pace maker or automatic defibrillator, implanted insulin pump
  * auditory neurostimulator, anal neurostimulator, etc.
  * ferromagnetic bodies in soft tissues, intraocular foreign bodies, cerebral vascular clips
  * claustrophobia
  * morphotype not allowing access to MRI: morbid obesity with waist circumference greater than 150 cm, shoulder width greater than 59 cm
* Patient with psychiatric pathology (untreated psychosis, drug dependence, etc.)
* Pregnant or breast-feeding patient
* Patient in periods of exclusion (determined by a previous or ongoing study)
* Patient under safeguard of justice
* Patient under guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Changes in body weight | Before preparation, before surgery, and at 1 month, 3 months, 6 months, 12 months and 24 months after surgery
  Changes in body weight
Excess weight loss | 2 years after surgery
  The percentage of excess weight loss is obtained as follow:
  (initial body weight - body weight at 2 years postoperatively) / (initial body weight - ideal body weight at BMI 25) x 100
Changes in Body Mass Index (BMI) | Before preparation, before surgery, and at 1 month, 3 months, 6 months, 12 months and 24 months after surgery
  Changes in Body Mass Index, obtained as follow:
  body weight (in kilograms)/ the square of height (in meters)

SECONDARY OUTCOMES:
Changes in the physical status in terms of muscle/fat report | Before preparation, before surgery and 24 months after surgery
  Muscle/ Fat Cross Sectional Area report obtained by the mean of Magnetic Resonance Imaging (MRI)
Changes in the physical status in terms of walking abilities | before preparation, before surgery, and at 1 month, 3 months, 6 months, 12 months and 24 months after surgery
  Changes in 6-min walk test: the distance (in meters) that the patient is able to walk in 6 minutes
Changes in the physical status in terms of waist circumference | before preparation, before surgery, and at 1 month, 3 months, 6 months, 12 months and 24 months after surgery
  Changes in waist circumference measured in centimetres
Changes in physical status in terms of hip circumference | before preparation, before surgery, and at 1 month, 3 months, 6 months, 12 months and 24 months after surgery
  Changes in hip circumference measured in centimetres
Changes in surgical difficulty in terms of left liver volume | Before preparation, before surgery and 24 months after surgery
  Left liver volume, as measured by Magnetic Resonance Imaging (MRI)
Changes in surgical difficulty in terms of visceral flat volume | Before preparation, before surgery and 24 months after surgery
  Visceral Fat volume, as measured by Magnetic Resonance Imaging (MRI) on a 1 cm slide at L2-L3 level
Comparison of surgical difficulty in terms of surgery duration | At time of surgery
  Total duration of Surgery, in minutes, for each group
Comparison of surgical difficulty in terms of gastric pouch positioning duration | At time of surgery
  Time from trocar positioning to fashioning the gastric pouch, in minutes, for each group
Comparison of surgical difficulty in terms of postoperative hospitalisation duration | At time of surgery
  Duration of the hospitalisation stay after the surgery, in days, for each group
Changes in the quality of life by the mean of the Gastrointestinal Quality of Life Index (GIQLI) | before preparation, before surgery, and at 1 month, 3 months, 6 months, 12 months and 24 months after surgery
  The GIQLI (Gastrointestinal Quality of Life Index) questionnaire is a digestive quality of life score including 36 items dealing with symptoms, physical status, emotions, social problems, and the effect of medical treatment in relation with gastro-intestinal disorders or procedures. The score is between 0 and 144, the higher the score, the better the quality of life.
Changes in the quality of life by the mean of a quality of life questionnaire specialized in bariatric surgery | before preparation, before surgery, and at 1 month, 3 months, 6 months, 12 months and 24 months after surgery
  "Moorehead-Ardelt Quality of Life Questionnaire II" (M-A-QoLQII) was originally designed as a disease-specific instrument to measure postoperative outcomes of self-perceived QoL in obese patients. Six areas are examined: self-esteem, physical well-being, social relationships, work, sexuality, and eating behavior. Each item is evaluated on a 10-point scale and scored from -0.5 to +0.5. The higher the score, the better the quality of life.
Changes in the remission rate of fatty liver | Before preparation, before surgery and 24 months after surgery
  the remission rate of the fatty liver is assessed by MRI (Magnetic Resonance Imaging) which provides measurements of the liver fatty infiltration
Changes in liver elasticity | Before preparation, before surgery and 24 months after surgery
  The liver elasticity is assessed by Magnetic Resonance Elastography (MRE) which provides quantitative maps of its stiffness
Changes in iron overload in the liver | Before preparation, before surgery and 24 months after surgery
  The iron overload in the liver is assessed through Magnetic Resonance Imaging (MRI) measurement of the tissue relaxivity in T2 phase
Changes in LDL cholesterol levels | Before preparation, before surgery and 24 months after surgery
  Changes in LDL cholesterol levels (grams per liter)
Changes in insulin resistance | Before preparation, before surgery and 24 months after surgery
  Changes in Homeostatic Model Assessment of Insulin Resistance(HOMA-IR) levels is calculated as follow:
  HOMA - IR = Insulin x Glucose / 22.5
Surgical complication assessment | Up to 24 months after surgery
  percentage of patients presenting a complication

CONTACTS AND LOCATIONS:
Overall Officials: Michel VIX, MD, PhD, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2985-3023. doi: 10.1016/j.jacc.2013.11.004. Epub 2013 Nov 12. No abstract available. PMID 24239920
- [Background] Yang YX, Chong MS, Lim WS, Tay L, Yew S, Yeo A, Tan CH. Validity of estimating muscle and fat volume from a single MRI section in older adults with sarcopenia and sarcopenic obesity. Clin Radiol. 2017 May;72(5):427.e9-427.e14. doi: 10.1016/j.crad.2016.12.011. Epub 2017 Jan 20. PMID 28117037
- [Background] Maislin G, Ahmed MM, Gooneratne N, Thorne-Fitzgerald M, Kim C, Teff K, Arnardottir ES, Benediktsdottir B, Einarsdottir H, Juliusson S, Pack AI, Gislason T, Schwab RJ. Single slice vs. volumetric MR assessment of visceral adipose tissue: reliability and validity among the overweight and obese. Obesity (Silver Spring). 2012 Oct;20(10):2124-32. doi: 10.1038/oby.2012.53. Epub 2012 Mar 7. PMID 22395811
- [Background] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697
- [Background] Moorehead MK, Ardelt-Gattinger E, Lechner H, Oria HE. The validation of the Moorehead-Ardelt Quality of Life Questionnaire II. Obes Surg. 2003 Oct;13(5):684-92. doi: 10.1381/096089203322509237. PMID 14627461
- See also: The ASMBS textbook of bariatric surgery — https://www.academia.edu/38470266/The_ASMBS_Textbook_of_Bariatric_Surgery_Vol